CLINICAL TRIAL: NCT06773923
Title: Effectiveness of Patient-specific 3D-printed Resorbable Scaffolds of Polycaprolactone, Beta-tricalcium Phosphate, and Metformin Used for Maxillary Bone Regeneration: Randomized Clinical Trial
Brief Title: Effectiveness of 3D-printed Patient-specific Resorbable Scaffolds for Maxillary Bone Regeneration
Acronym: OSTEOPRINT
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Austral de Chile (Other)
Responsible Party: Principal Investigator, Pedro C Aravena, DDS, PhD, Dental Implant and Periodontal Plastic Surgery Specialist, Universidad Austral de Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Osteoprint_2025; 23IRLR-249819 (Other Grant/Funding Number: Innova CORFO. Government of Chile)
Record Dates: First submitted 2025-01-07; First posted 2025-01-14 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Bone Loss; Jaw, Edentulous; Edentulous Mouth; Jaw Fractures; Bone Loss, Age Related
Keywords: Polycaprolactone; Scaffold; Bone regeneration; Printing, three dimensional; Dentistry; Clinical Trial
MeSH Terms: conditions — Bone Diseases, Metabolic; Jaw, Edentulous; Mouth, Edentulous; Jaw Fractures; Osteoporosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Osteoprint group (Experimental): Patients with of their jaw/jawbone in which the 3D scaffold printed with PCL will be inserted.
  Interventions: Device: PCL Scaffold
- Control group (Active Comparator): Patients with of their jaw/mandible which will be regenerated using the conventional technique using a titanium reinforced polytetrafluoroethylene (PTFE) membrane (Cytoplast® brand) and filling the space with Bio-Oss xenograft (Geistlich Pharma AG. Germany).
  Interventions: Device: PTFE + Bio-Oss®

INTERVENTIONS:
Device: PCL Scaffold — patients with their jaw/maxilla in which the 3D scaffold with PCL will be inserted.
  Arms: Osteoprint group
Device: PTFE + Bio-Oss® — patients with jaw/maxilla which will be regenerated using the conventional technique using a titanium reinforced polytetrafluoroethylene (PTFE) membrane (Cytoplast® brand) and filling the space with Bio-Oss xenograft (Geistlich
  Arms: Control group

SUMMARY:
The objective of this study is to test the bone formation capacity of a 3D printed scaffold with a plastic material called Polycaprolactone (PCL), compared to the use of synthetic bone grafts, for bone formation in the maxilla or mandible of elderly patients in the city of Valdivia between the years 2023-2024.

The main beneficiaries will be patients, users of the public or private health system, who require bone regeneration. The intermediate beneficiaries are the health team: doctors specializing in surgery and orthopedics, dentists, maxillofacial surgeons, dedicated to bone reconstruction and regeneration.

The innovation of this new material is based on the provision of a biocompatible plastic, easy to handle, for domestic 3D printing of bone matrices that can be grafted in areas requiring bone regeneration.

DETAILED DESCRIPTION:
A parallel-arm randomized clinical trial will be designed. The participants will be elderly patients from the city of Valdivia, Chile, regardless of sex, from the Dental Health Service of the Base Hospital of Valdivia for dental rehabilitation with dental implants. Clinical characteristics and complete medical history (such as sex, age and comorbidities) will be recorded and all the information that allows the identification of the patients will be encrypted.

Patients requiring bone regeneration at the time of examination should have an atrophic bilateral mandible with poor bone available according to periodontal diseases classification behind tooth #3.3 or #4.3; with an edentulous alveolar ridge with a remaining bone height of ≤ 6 mm. Patients will be excluded if they have had previous dental implant surgeries, with maxillary sinus pathologies, with oral tissue lesions, diseases that produce acute/chronic pain, smokers of more than 5 cigarettes per day, with excessive alcohol consumption (more than three times per week), and who suffer from any systemic disease whose surgical intervention is prohibited, for example: severe heart disease, congenital coagulation factor deficiency, dialysis, or malignant tumor in terminal phase. Also excluded are patients with diabetes that is not well controlled or who have difficulty achieving an Hb ≥ 7 g/dL in a preoperative examination; patients taking any anti-platelet or anticoagulant drug and patients with a history of heart disease.

- Sample size calculation Considering as the main objective of this study the formation of vital and functional bone analyzed in histological specimens, for the sample calculation the researcher relied on the previously randomized clinical trial who demonstrated a difference in the percentage of bone formation using PCL bone matrices in bone preservation was 9.5%. As a result of using this effect size with a given alpha level of 0.05, a power of 80% and an allocation ratio of 1, the sample size was 4 patients per group (algorithm: mean power 1 9.5, sd(3.6). STATA v.14.0..

Furthermore, taking into account that each patient will use both sides of their jaw (left and right), with two study groups and a 25% loss to follow-up or sample processing error, estimating that a total of 10 patients will participate in this study.

* Study groups and randomization

  * Osteoprint group: Patients with a jaw/maxilla atrophy in which the 3D scaffold with PCL will be inserted.
  * Control group: Patients with a jaw/maxilla atrophy which will be regenerated using the conventional technique using a titanium reinforced polytetrafluoroethylene (PTFE) membrane (Cytoplast® brand) and filling the space with Bio-Oss xenograft (Geistlich Pharma Agency. Germany).
* Randomization: The mechanism to perform the randomization sequence will be using the "RANDBETWEEN" function of Microsoft Excel® v.15.24.2016 (Microsoft, Sacramento. USA). An researcher will randomize in a spreadsheet with three columns: the first column with the patient number, the second column with the maxilla/mandible side to be used (#1 right side; #2 left side) and the third column with the type of study group to be used (#1: experimental group; #2: control group). This sequence will be previously determined by an investigator and will be informed before surgery, according to the number of patients to be operated.
* Experimental Design To analyze the osteogenic capacity of the 3D printed bone scaffold with PCL, an researcher will compare the volume of bone formed in the area using the 3D printed bone scaffold with PCL+ βTCP (experimental group) versus the volume of bone regenerated using a titanium-reinforced polytetrafluoroethylene (PTFE) membrane (control group). The outcome will be measured in histomorphometry and immunohistochemistry of bone biopsies obtained at six months.

ELIGIBILITY:
Inclusion Criteria:

* patients from the city of Valdivia, Chile, from Dental Health Service of the Base Hospital of Valdivia for the rehabilitation of their teeth with dental implants,
* age between 30 and 70 years old,
* regardless of sex,
* complete medical history (such as sex, age and comorbidities) will be recorded.
* patients requiring bone regeneration at the time of examination should have an atrophic bilateral mandible with poor bone available according to periodontal deseases classification behind tooth #3.3 or #4.3; with an edentulous alveolar ridge with a remaining bone height of ≤ 6 mm.

Exclusion Criteria:

* patients had previous dental implant surgeries,
* with maxillary sinus pathologies or oral tissue lesions,
* diseases that produce acute/chronic pain,
* smokers of more than 5 cigarettes per day,
* with excessive alcohol consumption (more than three times per week),
* who suffer from any systemic disease whose surgical intervention is prohibited, for example: severe heart disease, congenital coagulation factor deficiency, dialysis, or malignant tumor in terminal phase,
* patients with diabetes that is not well controlled or who have difficulty achieving an Hb ≥ 7 g/dL in a preoperative examination,
* patients taking any antiplatelet or anticoagulant drug,
* patients with a history of heart disease.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Histology: area new bone tissue | 6 months
  Bone biopsies obtained during implant installation surgery will be used. Once mounted on slides and stained with hematoxylin-eosin (H&E) and immunohistochemical markers, they will show the presence of vital bone as bone tissue with osteocyte lacunae, soft connective tissue and blood vessels. The amount of new bone tissue will be quantified as the percentage of area encompassed by the new bone sample versus the field of view observed under the light microscope at 40X magnification.
Biomarkers | 6 months
  In bone biopsies with inmunohistochemistry markers, optical densities of interferon-α, IL-1β, interleukin -10 t Runx-2 positive stains as percentage of the total area observed in the microscope field will be registered.

SECONDARY OUTCOMES:
Oral Health Quality of life. | 6 months
  All patients will be given the "Health-related quality of life (HRQOL) scale in its Spanish version 'HRQOL-sp'. The scale evaluates symptoms, psychological aspects and oral function. This instrument is specifically used to measure patients' perception after surgery in four domains (oral function, general activity, signs and symptoms, and pain) and the recording of postoperative associated signs or symptoms, complications and pain level measured by the Verbal Rating Scale (VRS). The patients will be choice between four Likert scale alternatives: "no problems", "little problems", "quite a lot of problems" and "many problems".
Postoperative complications | 6 months
  The presence of dichotomous (yes/no) signs of: swelling, ecchymosis, bleeding, nausea, vomiting, fever will be quantified.
Level of pain | 6 months
  The level of pain felt during the follow-up between 1st to 14th day will be measured with a visual analog scale from 0 (no pain) to 10 points (worst pain imaginable).

CONTACTS AND LOCATIONS:
Locations (1):
- Valdivia, Valdivia, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dalfino S, Olaret E, Piazzoni M, Savadori P, Stancu I, Tartaglia G, Dolci C, Moroni L. Polycaprolactone/beta-Tricalcium Phosphate Composite Scaffolds with Advanced Pore Geometries Promote Human Mesenchymal Stromal Cells' Osteogenic Differentiation. Tissue Eng Part A. 2025 Jan;31(1-2):13-28. doi: 10.1089/ten.TEA.2024.0030. Epub 2024 Apr 30. PMID 38613813
- [Background] Rai B, Lin JL, Lim ZX, Guldberg RE, Hutmacher DW, Cool SM. Differences between in vitro viability and differentiation and in vivo bone-forming efficacy of human mesenchymal stem cells cultured on PCL-TCP scaffolds. Biomaterials. 2010 Nov;31(31):7960-70. doi: 10.1016/j.biomaterials.2010.07.001. Epub 2010 Aug 4. PMID 20688388
- [Background] Park H, Kim JS, Oh EJ, Kim TJ, Kim HM, Shim JH, Yoon WS, Huh JB, Moon SH, Kang SS, Chung HY. Effects of three-dimensionally printed polycaprolactone/beta-tricalcium phosphate scaffold on osteogenic differentiation of adipose tissue- and bone marrow-derived stem cells. Arch Craniofac Surg. 2018 Sep;19(3):181-189. doi: 10.7181/acfs.2018.01879. Epub 2018 Sep 20. PMID 30282427
- [Background] Safiaghdam H, Nokhbatolfoghahaei H, Farzad-Mohajeri S, Dehghan MM, Farajpour H, Aminianfar H, Bakhtiari Z, Jabbari Fakhr M, Hosseinzadeh S, Khojasteh A. 3D-printed MgO nanoparticle loaded polycaprolactone beta-tricalcium phosphate composite scaffold for bone tissue engineering applications: In-vitro and in-vivo evaluation. J Biomed Mater Res A. 2023 Mar;111(3):322-339. doi: 10.1002/jbm.a.37465. Epub 2022 Nov 5. PMID 36334300
- [Background] Rodrigues MT, Martins A, Dias IR, Viegas CA, Neves NM, Gomes ME, Reis RL. Synergistic effect of scaffold composition and dynamic culturing environment in multilayered systems for bone tissue engineering. J Tissue Eng Regen Med. 2012 Nov;6(10):e24-30. doi: 10.1002/term.499. Epub 2012 Mar 27. PMID 22451140
- [Background] Ivanovski S, Breik O, Carluccio D, Alayan J, Staples R, Vaquette C. 3D printing for bone regeneration: challenges and opportunities for achieving predictability. Periodontol 2000. 2023 Oct;93(1):358-384. doi: 10.1111/prd.12525. Epub 2023 Oct 12. PMID 37823472
- [Background] Obregon F, Vaquette C, Ivanovski S, Hutmacher DW, Bertassoni LE. Three-Dimensional Bioprinting for Regenerative Dentistry and Craniofacial Tissue Engineering. J Dent Res. 2015 Sep;94(9 Suppl):143S-52S. doi: 10.1177/0022034515588885. Epub 2015 Jun 29. PMID 26124216
- [Background] Ivanovski S, Staples R, Arora H, Vaquette C, Alayan J. Alveolar bone regeneration using a 3D-printed patient-specific resorbable scaffold for dental implant placement: A case report. Clin Oral Implants Res. 2024 Dec;35(12):1655-1668. doi: 10.1111/clr.14340. Epub 2024 Aug 7. PMID 39109582
- [Background] Park JY, Jeon SH, Lee JY, Park JM, Cha JK. Vertical and Horizontal Ridge Augmentation Using Customized Three-Dimensionally Printed Polycaprolactone Mesh in Atrophic Posterior Maxillae: A Case Report. J Oral Implantol. 2025 Aug 8;51(4):326-336. doi: 10.1563/aaid-joi-D-22-00007. PMID 36796059